CLINICAL TRIAL: NCT03186729
Title: Study of Antithrombotic Treatment After IntraCerebral Haemorrhage
Acronym: STATICH
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of resources
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Torgeir Bruun Wyller, Project leader, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Version/date 180315
Record Dates: First submitted 2017-06-08; First posted 2017-06-14 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Hemorrhage; Intracranial Hemorrhages; Atrial Fibrillation; Anticoagulant-Induced Bleeding; Secondary Prevention
Keywords: Intracerebral hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage; Intracranial Hemorrhages; Atrial Fibrillation | interventions — Fibrinolytic Agents

STUDY DESIGN:
Intervention Model Description: Randomised-controlled trial, parallel groups
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Antithrombotic treatment (Experimental): For patients with vascular disease and indication for antiplatelet drugs: Antiplatelet drugs; For patients with atrial fibrillation and indication for anticoagulant drugs: Anticoagulant drugs
  Interventions: Drug: Antithrombotic Agent
- No antithrombotic treatment (No Intervention): For patients with indication for antiplatelet drugs: No antithrombotic drugs For patients with atrial fibrillation and indication for anticoagulant drugs: No anticoagulant drugs.

INTERVENTIONS:
Drug: Antithrombotic Agent — Anticoagulant or antiplatelet drugs
  Arms: Antithrombotic treatment

SUMMARY:
The study evaluates the effects of antithrombotic drugs (anticoagulant drugs or antiplatelet drugs) for prevention of ischaemic events in patients With recent intracerebral haemorrhage.

DETAILED DESCRIPTION:
Patients with spontaneous ICH have an increased risk of recurrent ICH and they also have an increased risk of ischaemic diseases. Around 40-50% of patients use, or have an indication, for antithrombotic drugs at the time of ICH. However, little is known about the benefits and harms of using antithrombotic drugs for prevention of ischaemic events in patients who have had an ICH.

There are only observational studies addressing this question. Because of the lack of randomised-controlled trials and the inconclusive findings of the observational studies, guidelines have variably endorsed both starting and avoiding antithrombotic drugs after ICH.

The investigators therefore want to study the effect and safety of using antithrombotic drugs after ICH. Furthermore, since findings on MRI can be biomarkers for subsequent bleeding, there will also be performed a sub-study of the association between such findings on MRI and risk of recurrent ICH during treatment with antithrombotic drugs.

Patients with ICH during the last 6 months and with an indication for antithrombotic drugs will be included. Patients with vascular disease and indication for antiplatelet drugs will be randomised to antiplatelet treatment vs. no antithrombotic treatment. Patients with atrial fibrillation and indication for anticoagulant treatment will be randomised to anticoagulant treatment vs. no anticoagulant treatment. The follow up period is 2 years, and the primary effect variable is new ICH. The investigators will also assess new intracranial haemorrhage, extracranial haemorrhage and ischemic events, and functional and cognitive outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥18 years.
* Spontaneous, primary ICH, of ≥1 day, but not more than 180 days after onset of qualifying ICH, i.e.:

  * No preceding traumatic brain injury, based on history from the patient/witness of spontaneous symptom onset, and brain imaging appearances consistent of spontaneous ICH (i.e. any brain/bone/soft tissue appearances of trauma must have occurred secondary to a spontaneous ICH)
  * No 'secondary' or underlying structural cause (e.g. haemorrhagic transformation of an ischaemic stroke, aneurysm, tumour, arteriovenous malformation, or intracerebral venous thrombosis)
* Patient have indication for antithrombotic (i.e. anticoagulant or antiplatelet) drug for the prevention of ischaemic events, either antiplatelet drugs (for patients with vascular disease), or anticoagulant drug for patients with atrial fibrillation.
* Consent to randomisation from the patient (or personal / legal / professional representative if the patient does not have mental capacity).
* MRI (or CT) is performed before randomisation.

Exclusion Criteria:

* Clear indication for antiplatelet or anticoagulant treatment (e.g. prosthetic heart valves).
* Contraindications to the antithrombotic drug that will be administered.
* Patient is pregnant, breastfeeding, or of childbearing age and not taking contraception.
* For patients examined with MRI: Contraindication for brain MRI
* Malignancy with life expectancy less than 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Fatal or non-fatal symptomatic ICH. | 2 years
  Neurological deterioration or death associated with intracerebral haemorrhage found on CT scan, MRI, or autopsy.

SECONDARY OUTCOMES:
Functional outcome | 2 years
  Modified Rankin Scale score
Death of any cause | 2 years
  Death of any cause
Vascular death | 2 years
  Death of vascular cause
Symptomatic epidural, subdural, or subarachnoid haemorrhage | 2 years
  Neurological deterioration or death associated with epidural, subdural, or subarachnoid haemorrhage found on CT scan, MRI, or autopsy.
Symptomatic major extracranial haemorrhage | 2 years
  Clinically overt bleeding associated with one or more of:
  * Transfusion of >2 red cell units of blood
  * A fall in haemoglobin of 2 g/dL, (1.24 mmol/L)
  * Bleeding into retroperitoneum, intraocular space or major joint
  * Bleeding leading to permanent treatment cessation
Ischaemic events | 2 years
  Transient ischaemic attack, ischaemic stroke, unstable angina, acute myocardial infarction (type 1), peripheral arterial occlusion, mesenteric ischaemia, retinal arterial occlusion, deep vein thrombosis or pulmonary embolism.

CONTACTS AND LOCATIONS:
Overall Officials: Torgeir Bruun Wyller, PhD, Principal Investigator — Oslo University Hospital
Locations (3):
- Herlev Gentofte Hospital, Copenhagen, Denmark
- Oslo University Hospital, Oslo, Norway
- Umeå University Hospital, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared within the COCROACH Collaboration.

REFERENCES:
- [Derived] Li L, Poon MTC, Samarasekera NE, Perry LA, Moullaali TJ, Rodrigues MA, Loan JJM, Stephen J, Lerpiniere C, Tuna MA, Gutnikov SA, Kuker W, Silver LE, Al-Shahi Salman R, Rothwell PM. Risks of recurrent stroke and all serious vascular events after spontaneous intracerebral haemorrhage: pooled analyses of two population-based studies. Lancet Neurol. 2021 Jun;20(6):437-447. doi: 10.1016/S1474-4422(21)00075-2. PMID 34022170
- [Derived] Cheng X, Dong Q. Towards individualised secondary prevention after intracerebral haemorrhage. Lancet Neurol. 2021 Jun;20(6):411-413. doi: 10.1016/S1474-4422(21)00130-7. No abstract available. PMID 34022160

DOCUMENTS (2):
  • Study Protocol (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/29/NCT03186729/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-28): https://cdn.clinicaltrials.gov/large-docs/29/NCT03186729/SAP_001.pdf